CLINICAL TRIAL: NCT00564239
Title: Efficacy of Child-centered Cognitive-Behavioral Prevention of Internalizing Disorders and the Impact of Simultaneous Parent Training
Brief Title: Psychological Prevention of Internalizing Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Institute of Behavioral-Therapy and -Medicine at the Philipps University Marburg (Other); Dept. of Child and Adolescent Psychiatry, Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Jan Pauschardt, Dr. rer. nat., Philipps University Marburg
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IVV-001-2007; IVV-001-2007
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Anxiety Symptoms; Depressive Symptoms; Somatoform Symptoms
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Group Therapy
- B (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Group Therapy
- C (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Group Therapy — 12 children group sessions, 8 parent group sessions
  Arms: A
Behavioral: Cognitive Behavioral Group Therapy — 12 children group sessions
  Arms: B

SUMMARY:
The purpose of this study is to determine whether cognitive-behavioral group prevention (CBT-G) for german children is effective and to what extent parental group training moderates outcome.

DETAILED DESCRIPTION:
Internalizing disorders represent a large group of psychological disorders among children who are referred to psychological treatment. Anxiety, Depression and somatoform disorders in children and adolescents increase the risk of mental disorders in adulthood. Some english programs have proved the efficacy of CBT-G prevention.This study will test the efficacy of CBT-G in German children. The role of parental involvement is currently subject to scientific discussions. The impact of an additional parent-group training will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* age 8- 12 years and
* anxiety symptoms and/or
* depressive symptoms and/or
* somatoform symptoms

Exclusion Criteria:

* psychiatric disorder according to ICD-10/ DSM-IV-TR requiring individual psychotherapy
* IQ < 85

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist (german version) | 3, 6, 18 months

SECONDARY OUTCOMES:
Inventar zur Erfassung der Lebensqualität bei Kindern und Jugendlichen (ILK)- Assessment of life quality, parent and child versions | 3, 6, 18 months
Spence Children's Anxiety Scale (SCAS) | 3, 6, 18 months
Depressionsinventar für Kinder- und Jugendliche (DIKJ), german depression inventory based on CDI | 3, 6, 18 months
Giessener Beschwerdebogen für Kinder- und Jugendliche (GBB-KJ), report of somatic symptoms, parent and child versions | 3, 6, 18 months
Culture Fair Intelligence Test (CFT 20-R) | initially
Symptom-Checklist (SCL-90-R), german version | 3, 6, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Pauschardt, Dr., Principal Investigator — Philipps University Marburg; Sylvia D Eimecke, Dr., Principal Investigator — Philipps University Marburg; Fritz Mattejat, PhD, Study Director — Philipps University Marburg
Locations (1):
- Institut für Verhaltenstherapie und -medizin (IVV), Marburg, Hesse, Germany